CLINICAL TRIAL: NCT05642117
Title: Pediatric Telephone Center Board 15 and Adhesion Factors
Brief Title: Pediatric Telephone Center Board 15
Acronym: CTPC15
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: CTPC15 - 29BRC21.0124
Record Dates: First submitted 2021-05-10; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Emergencies; Pediatric ALL; Response, Acute Phase
Keywords: Urgent Medical Aid Service (SAMU); Pediatric
MeSH Terms: conditions — Emergencies; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Acute-Phase Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the follow-up of advices given in a Urgent Medical Aid Service (SAMU 29) for every pediatric's emergency call under 15yo and try to evaluate the adhesion's factors.

DETAILED DESCRIPTION:
Many of pediatric's medical emergency are followed by a medical advice in a Urgent Medical aid Service (SAMU).

This advices could be medications advices, to see a general praticionner the same day or later, or to consult in an emergency department.

But the rate of advices really followed by callers is unknown. This study evaluate by who, when and why this advices are followed or not.

ELIGIBILITY:
Inclusion Criteria:

* all emergency calls at SAMU 29 for under 15yo childs
* medical advices were given by the physician (medication at home OR consult in an emergency department OR consult the general praticionner the same day or later.

Exclusion Criteria:

* all emergency calls at SAMU 29 for upper 15yo childs
* participation opposition.
* need for an ambulance or an emergency medical team at home

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all pediatric's emergency call for a child Under 15yo with a medical advice given by the physician.
Sampling Method: Non-Probability Sample
Enrollment: 785 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
rate of medical advices with follow-up completed in epidemic condition | 10 days
  number of medical advices followed after calling SAMU in epidemic condition
rate of medical advices with follow-up completed in summer | 10 days
  number of medical advices followed after calling SAMU in summer

SECONDARY OUTCOMES:
epidemiology of pediatric's emergency calls in Urgent Medical Aid Service (SAMU 29) | 10 days in epidemic condition
  Who, when and why population calls for an pediatric's emergency probleme
epidemiology of pediatric's emergency calls in Urgent Medical Aid Service (SAMU 29) | 10 days in summer
  Who, when and why population calls for an pediatric's emergency probleme
adhesion factors to follow medical advice | 10 days in epidemic condition
  By who, when and why medical advices were not followed by callers
adhesion factors to follow medical advice | 10 days in summer
  By who, when and why medical advices were not followed by callers

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France